CLINICAL TRIAL: NCT04486495
Title: Minimal Invasive Axillary Staging and Treatment After Neoadjuvant Systemic Therapy in Node Positive Breast Cancer (MINIMAX): a Dutch Multicenter Observational Study to Gain Insight in Less and More Invasive Axillary Staging and Treatment in Relation to Oncologic Safety and Quality of Life to Develop Evidence-based Guidelines.
Brief Title: Minimal Invasive Axillary Staging and Treatment After Neoadjuvant Systemic Therapy in Node Positive Breast Cancer
Acronym: MINIMAX
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-12518
Record Dates: First submitted 2020-07-07; First posted 2020-07-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Lymph Node Metastases
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, the majority of clinically node positive (cN+) breast cancer patients is treated with neoadjuvant systemic therapy (NST). Axillary staging and treatment after NST in cN+ patients are areas of controversy. Patients with a pathological complete response (pCR) of the axillary lymph nodes are not expected to benefit from axillary lymph node dissection (ALND). Hence, less invasive axillary staging procedures are being introduced to avoid unnecessary ALND. However, evidence supporting the safety of replacing ALND by less invasive techniques in terms of oncologic safety and impact on quality of life (QoL) is lacking.

DETAILED DESCRIPTION:
The MINIMAX is a multicenter registry study that includes node positive breast cancer patients, who are treated with NST (chemotherapy and ± immunotherapy), in order to gain insight in the oncologic safety and impact on QoL of less and more invasive axillary staging and treatment strategies.

Patients who are included in this study will complete Patient Reported Outcome Measures (PROMs) at baseline (time of diagnosis), and 1 and 5 years after diagnosis to assess impact on QoL.

A database will be built by the Netherlands Cancer Registry. Data on patient-, tumor-, pre-NST staging-, post-NST staging- and treatment-characteristics will be retrieved from patients' records by trained data registrars of the Netherlands Comprehensive Cancer Organisation (IKNL) using electronic case report forms (eCRFs). Five-year survival and recurrence will be evaluated to determine oncologic safety.

The results will be incorporated in the national guidelines. In case of an equilibrium between less and more invasive strategies, the data of this study will at least be extremely suitable to be used in the shared decision making process.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with unilateral invasive breast cancer and cN1-3
* Pathologically proven positive axillary lymph node
* Planned to undergo neoadjuvant chemotherapy (± immunotherapy), followed by staging and treatment of the breast and axilla

Exclusion Criteria:

* Clinically node negative breast cancer before NST
* Bilateral invasive breast cancer
* Neoadjuvant endocrine therapy
* Distant metastases (including oligometastatic disease)
* History of invasive breast cancer
* Other malignancies, except for basal/squamous cell skin cancer, and in situ carcinoma of the cervix or breast
* Axillary surgery or radiotherapy before NST (this includes SLNB prior to NST)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with unilateral invasive breast cancer and cN1-3, with a minimum of one pathologically proven positive axillary lymph node, treatment with neoadjuvant chemotherapy (± immunotherapy), followed by staging and treatment of the breast and axilla.
Sampling Method: Non-Probability Sample
Enrollment: 549 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 5 years
  DFS is defined as the time interval between the date of diagnosis until the date that a patient survives without any signs or symptoms of the disease.
Breast cancer specific survival (BCSS) | 5 years
  BCSS is defined as the time interval between the date of diagnosis until death from the disease.
Overall survival (OS) | 5 years
  OS is defined as the time interval between the date of diagnosis until death from any cause.
Axillary recurrence rate (ARR) | 5 years
  ARR is defined as tumor recurrence and as residual tumor that became clinically apparent in the ipsilateral axillary lymph nodes (pathologically proven).
Quality of life, as measured by EQ-5D-5L | Baseline, and 1 and 5 years after baseline
  The EQ-5D-5L comprises a descriptive system questionnaire and a visual analogue scale (VAS). The descriptive system consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, participants choose one of 5 levels that best describes their health on that day (from 'no problem'= 1 to 'unable/extreme'= 5). The numbers chosen for the five dimensions are combined to give a 5 digit score (minimum score = 11111 maximum score = 55555). The VAS provides participant's rating of their health on a scale from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine').
Quality of life, as measured by Quality of Life Questionnaire Core 30 Items (QLQ-C30) and QLQ-BR23 | Baseline, and 1 and 5 years after baseline
  These questionnaires contain functional domains, global health status, and symptom scales. For functional domains and global health status, scores range from 0 to 100 with higher scores representing a better level of functioning. For symptoms scales, scores range from 0 to 100 with higher scores representing a greater degree of symptoms.
Quality of life, as measured by BREAST-Q, which includes the following domains: satisfaction with breasts, psychosocial well being, physical well being, sexual well being. | Baseline, and 1 and 5 years after baseline
  All domains are scored 0 to 100 points. Higher points represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Smidt, MD, PhD, Principal Investigator — Maastricht University Medical Center; Marie-Jeanne Vrancken Peeters, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Linetta Koppert, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (35):
- Netherlands (35):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Northwest Clinics, Alkmaar
  - The Netherlands Cancer Institute, Amsterdam
  - Gelre Hospital, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Red Cross Hospital, Beverwijk
  - Alexander Monro Hospital, Bilthoven
  - Amphia Hospital, Breda
  - Van Weel-Bethesda, Dirksland
  - Slingeland Hospital, Doetinchem
  - Albert Schweitzer Hospital, Dordrecht
  - Gelderse Vallei Hospital, Ede
  - Catharina Hospital, Eindhoven
  - Máxima Medical Center, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Martini Hospital, Groningen
  - Saxenburgh Medical Center, Hardenberg
  - Ziekenhuisgroep Twente, Hengelo
  - Tergooi Hospital, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Dijklander Hospital, Hoorn
  - Medical Center Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Alrijne Hospital, Leiderdorp
  - Haaglanden Medical Center, Leidschendam
  - Maastricht University Medical Center, Maastricht
  - Canisius Wilhelmina Hospital, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Spijkenisse Medical Center, Spijkenisse
  - ZorgSaam Hospital, Terneuzen
  - Diakonessenhuis, Utrecht
  - Isala Hospital, Zwolle

IPD SHARING:
Plan to Share IPD: No